CLINICAL TRIAL: NCT03749954
Title: Detachable String Magnetically Controlled Capsule Endoscopy for Detecting High-risk Varices in Compensated Advanced Chronic Liver Disease (CHESS1801): A Prospective Multicenter Study
Brief Title: Detachable String Magnetically Controlled Capsule Endoscopy for Detecting High-risk Varices in Compensated Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Beijing 302 Hospital (Other); Sir Run Run Shaw Hospital (Other); Zhujiang Hospital (Other); Shandong Provincial Hospital (Other Government); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Second Provincial General Hospital (Other); The Fifth Affiliated Hospital of Zunyi Medical College (Other); LanZhou University (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Changhai Hospital (Other); The Second Affiliated Hospital of Baotou Medical College (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Professor, LanZhou University
Other Study IDs: CHESS1801
Record Dates: First submitted 2018-11-17; First posted 2018-11-21 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Compensated Cirrhosis; Gastroesophageal Varices Bleeding
Keywords: Magnetically controlled capsule endoscopy; Gastroesophageal varices bleeding; Varices needing treatment
MeSH Terms: interventions — Endoscopy; Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall eligible participants: Eligible participants will receive standard esophagogastroduodenoscopy and magnetically controlled capsule endoscopy (Ankon Medical Technologies Co. Ltd.).
  Interventions: Diagnostic Test: Detachable string magnetically controlled capsule endoscopy

INTERVENTIONS:
Diagnostic Test: Detachable string magnetically controlled capsule endoscopy — Esophagogastroduodenoscopy is performed 2 hours after the magnetically controlled capsule endoscopy (Ankon Medical Technologies Co. Ltd.).
  Other Names: Esophagogastroduodenoscopy

SUMMARY:
Gastroesophageal varices is a serious complication of compensated advanced chronic liver disease (cACLD). Primary prophylaxis to reduce the risk of variceal haemorrhage is recommended if high-risk varices (HRV) are detected. We performed this study to compare the accuracy, patients' satisfaction and safety of detection of HRV by detachable string magnetically controlled capsule endoscopy (DS-MCCE) with esophagogastroduodenoscopy (EGD) as the standard.

DETAILED DESCRIPTION:
The presence of gastroesophageal varices (GEV) is a common and serious complication of compensated advanced chronic liver disease (cACLD).1-3 GEV hemorrhage is associated with a six week mortality rate of between 15% and 25%.2,3 In order to prevent variceal hemorrhage, screening and surveillance aims to detect high-risk varices (HRV) and determine the need for primary preventative therapy.2,3 Esophagogastroduodenoscopy (EGD) is therefore an important part of the diagnostic work-up in patients with cACLD, serving as the gold standard to diagnose HRV.2,3 However, EGD is invasive and poorly tolerated, with many patients needing intravenous sedatives or general anesthesia. Although EGD with sedation relieves patients' anxiety and discomfort and reduces the potential for physical injury during the procedure, it incurs additional risks of cardiopulmonary adverse events.4 Consequently, patients may decline a screening procedure if they are stable and asymptomatic.

Non-invasive methods for detection of cACLD are being explored.5-13 Although preliminary research is encouraging, these techniques predict the presence, rather than confirm or assess the size, of GEV. By contrast, capsule endoscopy is a non-invasive alternative which also allows direct visualization of GEV.14 A number of well-conducted trials15-19 suggest that EGD and capsule endoscopy may be equivalent in terms of accuracy in the identification and grading of varices. However, concerns remain that the quality of examination may be adversely affected by the uncontrolled and sometimes rapid transit of the capsule through the esophagus.20 String capsule endoscopy was introduced to address this concern by providing control of capsule movement as well as real-time visualization.21 However, this technique is limited by the inability to detach the string from the capsule. Thus, observation of the fundus, one of the predilection sites of varices, is impossible and retrieval of the capsule from the esophagus causes discomfort.

Magnetically controlled capsule endoscopy (MCCE), a novel modality, was developed and approved by the China Food and Drug Administration in 2013.22 Our previous studies initially demonstrated that MCCE was comparable in accuracy to EGD for gastric examination.22,23 Furthermore, it has several strengths including non-invasiveness, no sedation requirement, and easy operation.22,23 We have since combined an innovative detachable string system with the MCCE (detachable string magnetically controlled capsule endoscopy (DS-MCCE)) and carried out a pilot study showing that DS-MCCE was safe and feasible both in healthy volunteers and patients with suspected esophageal disease.24 Moreover, successful detachment of the capsule from the string avoids the discomfort of retrieving the entire capsule from the mouth and allows subsequent investigation of the gastric cardia and fundus. To our knowledge, the diagnostic accuracy of HRV, comfort and safety of DS-MCCE in patients with cACLD have not been explored in a large-scale trial. This prospective, multicenter study aimed to assess the accuracy, patient's satisfaction, and safety of DS-MCCE for detecting HRV in well-characterized patients with cACLD.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years;
* confirmed cirrhosis based on liver biopsy or clinical findings;
* compensated cirrhosis;
* scheduled to undergo esophagogastroduodenoscopy;
* estimated survival time> 24 months, and model for end-stage liver disease (MELD) score< 19;
* with written informed consent.

Exclusion Criteria:

* contradictions for capsule endoscopy;
* contradictions for standard magnetic resonance imaging examination such as the presence of surgical metallic devices;
* pregnancy or unknown pregnancy status.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with compensated cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2022-11-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of magnetically controlled capsule endoscopy for the risk of variceal bleeding | 1 day
  Diagnostic accuracy of magnetically controlled capsule endoscopy to determine the high-risk or low-risk of variceal bleeding when compared with esophagogastroduodenoscopy as the reference standard

SECONDARY OUTCOMES:
Diagnostic accuracy of magnetically controlled capsule endoscopy for decompensation or death | 3 year
  Diagnostic accuracy of magnetically controlled capsule endoscopy to determine the presence or absence of decompensation (defined as development of ascites, bleeding, or overt encephalopathy) or death within 3-year follow-up
Diagnostic accuracy of other non-invasive methods for the risk of variceal bleeding | 1 day
  Diagnostic accuracy of other non-invasive methods to determine the high-risk or low-risk of variceal bleeding when compared with esophagogastroduodenoscopy as the reference standard
Diagnostic accuracy of other non-invasive methods for decompensation or death | 3 year
  Diagnostic accuracy of other non-invasive methods to determine the presence or absence of decompensation (defined as development of ascites, bleeding, or overt encephalopathy) or death within 3-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, M.D., Principal Investigator — LanZhou University
Locations (13):
- China (12):
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Zunyi Medical University, Zhuhai, Guangdong
  - Shandong Provincial Hospital affiliated to Shandong University, Jinan, Shandong
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Baotou Medical College, Baotou
  - Third Affiliated Hospital of Sun Yat-sen University, Guangzhou
- Sheffield Teaching Hospitals NHS Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] Liu F, Ning Z, Liu Y, Liu D, Tian J, Luo H, An W, Huang Y, Zou J, Liu C, Liu C, Wang L, Liu Z, Qi R, Zuo C, Zhang Q, Wang J, Zhao D, Duan Y, Peng B, Qi X, Zhang Y, Yang Y, Hou J, Dong J, Li Z, Ding H, Zhang Y, Qi X. Development and validation of a radiomics signature for clinically significant portal hypertension in cirrhosis (CHESS1701): a prospective multicenter study. EBioMedicine. 2018 Oct;36:151-158. doi: 10.1016/j.ebiom.2018.09.023. Epub 2018 Sep 27. PMID 30268833
- [Background] Qi X, Li Z, Huang J, Zhu Y, Liu H, Zhou F, Liu C, Xiao C, Dong J, Zhao Y, Xu M, Xing S, Xu W, Yang C. Virtual portal pressure gradient from anatomic CT angiography. Gut. 2015 Jun;64(6):1004-5. doi: 10.1136/gutjnl-2014-308543. Epub 2014 Nov 14. No abstract available. PMID 25398771
- [Background] Wang FS, Fan JG, Zhang Z, Gao B, Wang HY. The global burden of liver disease: the major impact of China. Hepatology. 2014 Dec;60(6):2099-108. doi: 10.1002/hep.27406. Epub 2014 Oct 29. PMID 25164003
- [Background] Zou WB, Hou XH, Xin L, Liu J, Bo LM, Yu GY, Liao Z, Li ZS. Magnetic-controlled capsule endoscopy vs. gastroscopy for gastric diseases: a two-center self-controlled comparative trial. Endoscopy. 2015 Jun;47(6):525-8. doi: 10.1055/s-0034-1391123. Epub 2015 Jan 15. PMID 25590177
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Berzigotti A, Seijo S, Arena U, Abraldes JG, Vizzutti F, Garcia-Pagan JC, Pinzani M, Bosch J. Elastography, spleen size, and platelet count identify portal hypertension in patients with compensated cirrhosis. Gastroenterology. 2013 Jan;144(1):102-111.e1. doi: 10.1053/j.gastro.2012.10.001. Epub 2012 Oct 8. PMID 23058320
- [Background] Bhardwaj A, Kedarisetty CK, Vashishtha C, Bhadoria AS, Jindal A, Kumar G, Choudhary A, Shasthry SM, Maiwall R, Kumar M, Bhatia V, Sarin SK. Carvedilol delays the progression of small oesophageal varices in patients with cirrhosis: a randomised placebo-controlled trial. Gut. 2017 Oct;66(10):1838-1843. doi: 10.1136/gutjnl-2016-311735. Epub 2016 Jun 13. PMID 27298379
- [Background] Rey JF, Ogata H, Hosoe N, Ohtsuka K, Ogata N, Ikeda K, Aihara H, Pangtay I, Hibi T, Kudo SE, Tajiri H. Blinded nonrandomized comparative study of gastric examination with a magnetically guided capsule endoscope and standard videoendoscope. Gastrointest Endosc. 2012 Feb;75(2):373-81. doi: 10.1016/j.gie.2011.09.030. Epub 2011 Dec 9. PMID 22154417
- [Derived] Wang S, Huang Y, Hu W, Mao H, McAlindon ME, Liu Y, Yang L, Zhang C, Xu M, He C, Dang T, Wu B, Ji D, Zhang L, Mao X, Zhang L, Liu C, Xu D, Li Y, Li G, Han J, Lv F, Liang X, Jin S, Zhang S, Tai FWD, Xu Q, Yang C, Wang G, Wang L, Li B, Yang H, Xie P, Deng L, Ren L, Chang Z, Wang X, Wang S, Gao X, Li J, Zhu L, Wang F, Zhang L, Zhang G, Jiang X, Pan J, Meng W, Li X, Hou J, Dray X, Liao Z, Qi X. Detachable string magnetically controlled capsule endoscopy for detecting high-risk varices in compensated advanced chronic liver disease (CHESS1801): A prospective multicenter study. Lancet Reg Health West Pac. 2020 Dec 11;6:100072. doi: 10.1016/j.lanwpc.2020.100072. eCollection 2021 Jan. PMID 34327406
- [Derived] Huang Y, Huang F, Yang L, Hu W, Liu Y, Lin Z, Meng X, Zeng M, He C, Xu Q, Xie G, Liu C, Liang M, Li X, Kang N, Xu D, Wang J, Zhang L, Mao X, Yang C, Xu M, Qi X, Mao H. Development and validation of a radiomics signature as a non-invasive complementary predictor of gastroesophageal varices and high-risk varices in compensated advanced chronic liver disease: A multicenter study. J Gastroenterol Hepatol. 2021 Jun;36(6):1562-1570. doi: 10.1111/jgh.15306. Epub 2020 Nov 18. PMID 33074566